CLINICAL TRIAL: NCT02601391
Title: Adapting the Systems Training and Emotional Predictability and Problem Solving Group (STEPPS) for Service Users With Complex Needs. A Pilot Evaluation of STEPPS High Intensity (STEPPS HI) Within Forensic Inpatient Services
Brief Title: An Evaluation of an Adapted STEPPS Group Within Forensic Services
Acronym: STEPPS-HI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to run research in the service. Research terminated.
Sponsor: Sussex Partnership NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Liz Collins, Trainee Forensic Psychologist, Sussex Partnership NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPFT-1
Record Dates: First submitted 2015-10-26; First posted 2015-11-10 (Estimated); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Personality Disorder
Keywords: STEPPS-HI; personality disorder; evaluation; forensic
MeSH Terms: conditions — Personality Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STEPPS within forensic services. (Other): Forensic inpatients attend the STEPPS-HI group. Consent will be obtained. Pre and post group psychometric questionnaires will be completed as well as each service user attending a short semi-structured interview following the conclusion of the group .
  Primary nurse will fill in pre and post group questionnaires. Facilitators will complete short feedback forms each session and attend a focus group upon completion.
  Psychology Assistants/Interns will collect records of self harm and violence/aggressive incidents for each service user as well as records of nursing observation level and leave status taken.
  Interventions: Behavioral: Adapting STEPPS within forensic inpatient services.

INTERVENTIONS:
Behavioral: Adapting STEPPS within forensic inpatient services. — This study will focus upon delivering the STEPPs-HI group within Forensic Healthcare Inpatient Services.
  Other Names: STEPPS-HI

SUMMARY:
The purpose of this study is to determine how effective the STEPPS-HI group is at improving emotional regulation skills in those with identified difficulties in this area within forensic inpatient services. In addition, to explore whether there is increased acceptability of the adapted STEPPS group (STEPPS-HI) for this client group.

DETAILED DESCRIPTION:
Systems Training for Emotional Predictability and Problem Solving (STEPPS) is a manualised group programme for people primarily with a diagnosis of Borderline Personality Disorder (BPD). Although, STEPPS groups have been run within prisons in USA, it has been less formally evaluated within forensic psychiatric settings except for Pipon-Young & Cole (2012). Taking the learning from these studies into account, significant adaptations to the current STEPPS manual are needed to increase the acceptability and applicability of the group within forensic settings.

Following the adaption of the STEPPS manual for a forensic inpatient population (STEPPS HI), this research aims to investigate how effective the group is at improving emotional regulation skills in those with identified difficulties in the area as well as whether there is increased acceptability of the adapted group for the participants. The outcome of the research is intended to provide feedback on the adaption of the STEPPS manual and also an evaluation of the revised programme.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* To give informed consent to participate in the study.
* Currently a resident in a low or medium secure unit.
* Has been diagnosed as meeting DSM-IV criteria for a personality disorder at some stage in their mental health history.
* Has identified difficulties with emotional regulation.
* Be willing and have suitable abilities to participate in a group.
* To be assessed by the clinical team as sufficiently psychologically robust to participate in the group and the research.

Exclusion Criteria:

* Psychiatric/psychological or any other difficulties that would mean that participants could not give informed consent.
* Intellectual/cognitive impairment which prohibits participants ability to consent or fully comprehend the study or study materials.
* Non-English speakers as there is no provision for interpreters.
* Unable to manage a group environment due to risk to self and others including bullying and violence (this will be assessed by the clinical and STEPPS-HI facilitation team.
* No evidence of emotional regulation difficulties.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
To assess change from baseline (start of group) on the Symptom Checklist-Revised (SCL-90-R), reassessing at end of group (26 weeks later). | Assess at baseline (start of group) and reassess end of group (26 weeks later)
  To assess change from baseline (start of group) on the Symptom Checklist-Revised (SCL-90-R), reassessing at end of group (26 weeks later).
To assess change from baseline (start of group) on the Zanarini Rating Scale for Borderline Personality Disorder, reassessing at end of group (26 weeks later). | Assess at baseline (start of group) and reassess end of group (26 weeks later)
  To assess change from baseline (start of group) on the Zanarini Rating Scale

SECONDARY OUTCOMES:
Modified Overt Aggression Scale (MOAS: Yudofsky, J. M. Silver, W. Jackson, J. Endicott, & D. W. Williams, 1986). | Assess at baseline (start of group) and reassess end of group (26 weeks later)
  Modified Overt Aggression Scale (MOAS: Yudofsky, J. M. Silver, W. Jackson, J. Endicott, & D. W. Williams, 1986).
Circumplex of Interpersonal Relationships in Closed Living Environments (CIRCLE; Blackburn & Renwick, 1996). | Assess at baseline (start of group) and reassess end of group (26 weeks later)
  Circumplex of Interpersonal Relationships in Closed Living Environments

OTHER OUTCOMES:
Number of self-harm incidents as assessed by Sussex Partnership NHS Foundation Trust Incident Reporting System. | A record of self-harm incidents will be collected weekly from one month prior to the group starting, weekly through the group intervention (26 weeks) and then weekly for one month after the group has finished (at 30 weeks).
  Data will be reviewed via assessing the Sussex Partnership NHS Foundation Trust Incident Reporting System. Key information will be extracted i.e. number of self-harm incidents within the time frames stated in the time frame section. An excel spread sheet to collect this information will be developed by the study's principal investigator and the data will be inputted into the spread sheet by the Psychology Interns. Data analysis (a paired-samples t-test) will be conducted to compare the mean rates of self-harm incidents pre-group and post group.
Number of violent incidents as assessed by Sussex Partnership NHS Foundation Trust Incident Reporting System. | A record of violent incidents will be collected weekly from one month prior to the group starting, weekly through the group intervention (26 weeks) and then weekly for one month after the group has finished (at 30 weeks).
  Data will be reviewed via assessing the Sussex Partnership NHS Foundation Trust Incident Reporting System. Key information will be extracted i.e. number of violent incidents within the time frames stated in the time frame section. An excel spread sheet to collect this information will be developed by the study's principal investigator and the data will be inputted into the spread sheet by the Psychology Interns. Data analysis (a paired-samples t-test) will be conducted to compare the mean rates of violent incidents pre-group and post group.
Assessing research participants (service users) views regarding group content, via attendance at a semi-structured interview utilising thematic analysis to analyse the data gathered (Braun & Clarke, 2006). | This will be completed at the end of the group intervention (26 weeks) with service users being invited to attend a semi-structured interview.
  Research participants will be invited to attend a 1-1 semi-structured interview to capture their views on group content, format, structure, process, non-attendance and drop-put rates. The qualitative data gathered will be analysed by the principal investigator using thematic analysis (Braun & Clarke, 2006).
Assessing research participants (group facilitators) views of the adapted group manual via attendance at a focus group, utilising thematic analysis to analyse the data gathered (Braun & Clarke, 2006). | This will be completed at the end of the group intervention (26 weeks) with group facilitators being invited to attend a focus group.
  Research participants will be invited to attend a focus group to capture overall views on the adapted manual. The qualitative data gathered will be analysed by the principal investigator using thematic analysis (Braun & Clarke, 2006).
Record of research participants (service users) observational levels as assessed by Sussex Partnership NHS Foundation Trust general, intermittent and within eyesight recording forms. | A record of observational level forms (general, intermittent and within eyesight) will be collected weekly from one month prior to group starting, weekly through group intervention (26 weeks) and then weekly for one month after the group has finished (at
  Data will be reviewed via assessing the Sussex Partnership NHS Foundation Trust record of observational level forms (general, intermittent and within eyesight). Key information will be extracted i.e. changes within observational levels in the time frames stated in the time frame section. An excel spread sheet to collect this information will be developed by the study's principal investigator and the data will be inputted into the spread sheet by the Psychology Interns. The data gathered will be reported in the demographic section of the result within the journal article developed to disseminate the outcomes of the study.
Record of leave status for each research participants (service user) as assessed by Sussex Partnership NHS Foundation Trust Mental Health Act 1983 - Section 17 Leave of Absence Forms. | A record of leave status will be collected weekly from one month prior to group starting, weekly through group intervention (26 weeks) and then weekly for one month after the group has finished (at 30 weeks).
  Data will be reviewed via assessing Sussex Partnership NHS Foundation Trust Mental Health Act 1983 - Section 17 Leave of Absence Forms for each research participant. Key information will be extracted i.e. changes within level status in the time frames stated in the time frame section. An excel spread sheet to collect this information will be developed by the study's principal investigator and the data will be inputted into the spread sheet by the Psychology Interns. The data gathered will be reported in the demographic section of the result within the journal article developed to disseminate the outcomes of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Collins, Principal Investigator — Sussex Partnership NHS Foundation Trust
Locations (1):
- Elizabeth Collins, Hellingly, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Black DW, Blum N, McCormick B, Allen J. Systems Training for Emotional Predictability and Problem Solving (STEPPS) group treatment for offenders with borderline personality disorder. J Nerv Ment Dis. 2013 Feb;201(2):124-9. doi: 10.1097/NMD.0b013e31827f6435. PMID 23364121
- [Background] Blackburn, R., & Renwick, S. J. (1996). Rating scales for measuring the interpersonal circle in forensic psychiatric patients. Psychological Assessment, 8, 76-84
- [Background] Blum, N., Bartels N., St. John, D., Pfohl, B. (2002). STEPPS: Systems Training for Emotional Predictability and Problem Solving: Group Treatment for Borderline Personality Disorder. Coralville, Iowa, Blum's Books.
- [Background] Braun, V. & Clarke, V. (2006). Using thematic analysis in psychology. Qualitative Research in Psychology, 3, 77 - 101.
- [Background] Connell, J. & Barkham, M. (2007). Core-10 User Manual, Version 1.1. Core System Trust & Core Information Management Systems Ltd.
- [Background] Dickinson T, Wright KM. Stress and burnout in forensic mental health nursing: a literature review. Br J Nurs. 2008 Jan 24-Feb 13;17(2):82-7. doi: 10.12968/bjon.2008.17.2.28133. PMID 18414278
- [Background] Gratz, K. L. & Roemer, E. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment, 26, 41-54.
- [Background] Harvey R, Black DW, Blum N (2010) STEPPS (Systems Training for Emotional Predictability and Problem Solving) in the United Kingdom: A preliminary report. Journal of Contemporary Psychotherapy. 40, 225-232.
- [Background] Pipon-Young, L., & Cole, S. (2012). A preliminary evaluation of the Systems Training for Emotional Predictability and Problem Solving (STEPPS) group in a women's forensic medium secure unit. Clinical Psychology Forum, 239, 35 - 39.
- [Background] Sarkar, J., & di Lustro, M. (2011). Evolution of secure services for women in England. Advances in Psychiatric Treatment, 17, 323-331.
- [Background] Yudofsky SC, Silver JM, Jackson W, Endicott J, Williams D. The Overt Aggression Scale for the objective rating of verbal and physical aggression. Am J Psychiatry. 1986 Jan;143(1):35-9. doi: 10.1176/ajp.143.1.35. PMID 3942284
- [Background] Zanarini MC, Vujanovic AA, Parachini EA, Boulanger JL, Frankenburg FR, Hennen J. Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD): a continuous measure of DSM-IV borderline psychopathology. J Pers Disord. 2003 Jun;17(3):233-42. doi: 10.1521/pedi.17.3.233.22147. PMID 12839102